CLINICAL TRIAL: NCT01230203
Title: Computed Tomography Scan Versus Color Duplex Ultrasound for Surveillance of Endovascular Repair of Abdominal Aortic Aneurysm. A Prospective Multicenter Study
Acronym: ESSEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-APN-01
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Endovascular Repair of Abdominal Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computed tomography scan versus color duplex ultrasound (Other)
  Interventions: Procedure: Computed tomography scan versus color duplex ultrasound

INTERVENTIONS:
Procedure: Computed tomography scan versus color duplex ultrasound — Computed tomography scan versus color duplex ultrasound

SUMMARY:
Cumulative radiation dose, cost, contrast induced nephrotoxicity and increased demand for computed tomography aortography (CTA) suggest that duplex ultrasonoraphy (DU) may be an alternative to CTA-based surveillance. The investigators compared CTA with DU during endovascular aneurysm repair (EVAR) follow-up.

Patients undergoing EVAR have radiological follow-up data entered in a prospectively multicenter database. The gold standard test for endoleak detection was CTA. DU interpretation was performed independently of CTA and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were followed after EVAR, whatever the trademark and the model of the stentgraft (bi-iliac or mono-iliac)
* Age > 18 years old
* Patient with social insurance
* Signature of informed consent

Exclusion Criteria:

* patients who underwent EVAR with a fenestrated or branched stentgraft
* Obese patients (BMI > 30)
* Patients with severe renal insufficiency (Creatinine Clearance < 30 ml/mn)
* Patients who can't practice both an CT scan with iode injection and duplex ultrasound test over a period of one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2010-12-16 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2015-06-12 (Actual)

PRIMARY OUTCOMES:
Clinically significant abnormalities that require secondary intervention (coil embolization, endovascular intervention, surgical conversion) | Between 1 week and 1 month
  Clinically significant abnormalities that require secondary intervention (coil embolization, endovascular intervention, surgical conversion) :
  * increasing aneurysm sac size (≥5mm),
  * type I or type III endoleak,
  * type II endoleak with an increasing aneurysm sac size (≥2mm)
  * significant stenosis of a limb of the stentgraft (≥70%).

SECONDARY OUTCOMES:
All abnormalities, clinically significant or no | Between 1 week and 1 month
  All abnormalities, clinically significant or no:
  All types of endoleak An increasing aneurysm sac size (≥1mm) Stenosis or thrombosis of limb of the stentgraft

CONTACTS AND LOCATIONS:
Overall Officials: Hassen-Khofja Reda, Principal Investigator — CHU de Nice - Service de Chirurgie Vasculaire
Locations (21):
- France (21):
  - CHU d'Amiens - Service de Chirurgie Vasculaire, Amiens
  - CHU d'Angers - Service de Chirurgie Vasculaire, Angers
  - CHU de Besançon - Service de Chirurgie Vasculaire, Besançon
  - CHU de Bordeaux - Service de Chirurgie Vasculaire, Bordeaux
  - CHU de Caen - Service de Chirurgie Vasculaire, Caen
  - CHU Clermont-ferrand - Service de Chirurgie Vasculaire, Clermont-Ferrand
  - AP-HP Créteil - Service de chirurgie vasculaire, Créteil
  - CHU de Dijon - Service de Chirurgie Vasculaire, Dijon
  - CHU de Grenoble - Service de Chirurgie Vasculaire, Grenoble
  - CHRU Lille Service de Chirurgie Vasculaire, Lille
  - HCL - Service de Chirurgie Vasculaire, Lyon
  - AP-HM Service de Chirurgie vasculaire, Marseille
  - APHM - Hôpital Nord - Service de Chirurgie Vasculaire, Marseille
  - CHU de Montpellier - Service de Chirurgie Vasculaire, Montpellier
  - CHU de Nantes - Service de Chirurgie Vasculaire, Nantes
  - CHU de Nice - Service de chirurgie vasculaire, Nice
  - AP-HP - Pitié Salpétrière - Service de Chirurgie Vasculaire, Paris
  - CHU de Rouen - Service de Chirurgie Vasculaire, Rouen
  - CHU de St Etienne - Service de Chirurgie Vasculaire, Saint-Etienne
  - CHU de Strasbourg - Service de Chirurgie Vasculaire, Strasbourg
  - CHU de Toulouse - Service de Chirurgie Vasculaire, Toulouse

REFERENCES:
- [Derived] Jean-Baptiste E, Feugier P, Cruzel C, Sarlon-Bartoli G, Reix T, Steinmetz E, Chaufour X, Chavent B, Salomon du Mont L, Ejargue M, Maurel B, Spear R, Midy D, Thaveau F, Desgranges P, Rosset E, Hassen-Khodja R; Association Universitaire de Recherche en Chirurgie Vasculaire. Computed Tomography-Aortography Versus Color-Duplex Ultrasound for Surveillance of Endovascular Abdominal Aortic Aneurysm Repair: A Prospective Multicenter Diagnostic-Accuracy Study (the ESSEA Trial). Circ Cardiovasc Imaging. 2020 Jun;13(6):e009886. doi: 10.1161/CIRCIMAGING.119.009886. Epub 2020 Jun 8. PMID 32507018